CLINICAL TRIAL: NCT05871827
Title: The Use of Intraoperative Fluoroscopic Computer Navigation on Hip Arthroplasty Component Position
Brief Title: THA With and Without Computer Navigation
Status: Completed | Type: Observational
Sponsor: Southeast Orthopedic Specialists (Network)
Responsible Party: Sponsor
Other Study IDs: DPS-JMP-2019-078
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hip Osteoarthritis; Avascular Necrosis of Hip
Keywords: total hip arthroplasty, computer navigation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional Overlay: Subjects who underwent THA without use of computer navigation
- Computer Navigation: Subjects who underwent THA with use of computer navigation
  Interventions: Procedure: Intraoperative Fluoroscopic Computer Navigation

INTERVENTIONS:
Procedure: Intraoperative Fluoroscopic Computer Navigation — Computer technology used during surgery
  Groups: Computer Navigation

SUMMARY:
The goal of this observational study is to compare postoperative results between patients who had total hip arthroplasty (THA) with and without the use of a computer navigation program. The main questions this study aims to answer are:

* Can using computer navigation produce better THA implant placement?
* Can using computer navigation make surgery more efficient?

Participant data collected include their postoperative x-rays and total operative time.

DETAILED DESCRIPTION:
The goal of this retrospective study is to compare implant placement and operative time of patients who underwent direct anterior total hip arthroplasty with and without the use of a computer navigation program. X-rays are used to measure acetabular cup orientation, leg length discrepancy, and total operative time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Direct Anterior (DA) THA with the principal investigator between August 2018 and February 2020 and received ACTIS stem and PINNACLE cup with or without computer navigation

Exclusion Criteria:

* Patients who underwent subsequent revision THA, conversion arthroplasty, hybrid procedures, experienced native or postoperative dislocations, and missing or inadequate radiographs at time of data collection.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent DA THA with the principal investigator between August 2018 and February 2020 and received ACTIS stem and PINNACLE cup.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Cup inclination | 12 weeks post op
  Acetabular cup orientation
Cup anteversion | 12 weeks post op
  Acetabular cup anteversion
Leg length discrepancy | 12 weeks post op
  Leg length discrepancy
Operative time | Immediate post op
  Operative time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: John Redmond, MD, Principal Investigator — Southeast Orthopedic Specialists
Locations (1):
- Southeast Orthopedic Specialists, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No